CLINICAL TRIAL: NCT05152563
Title: A Phase 3 Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacodynamic Effect of Subcutaneous AK002 in Subjects With Moderate to Severe Eosinophilic Gastritis and/or Eosinophilic Duodenitis
Brief Title: A Study to Assess Subcutaneous AK002 in Eosinophilic Gastritis and/or Eosinophilic Duodenitis
Acronym: ENIGMA-SC
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision
Sponsor: Allakos Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK002-023
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Eosinophilic Gastritis; Eosinophilic Duodenitis
Keywords: Eosinophil; Eosinophilic; Eosinophilic gastrointestinal disorders; EGID; EG; EGE; Eosinophilic Gastritis; Eosinophilic Duodenitis; Eosinophilic Gastroenteritis; EoD
MeSH Terms: conditions — Eosinophilic enteropathy; Eosinophilic Esophagitis | interventions — AK002

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SC 150 mg of lirentelimab (AK002) (Experimental): Subjects in this arm will receive 6 monthly doses of 150 mg of lirentelimab (AK002) administered subcutaneously.
  Interventions: Drug: AK002
- SC 300 mg of lirentelimab (AK002) (Experimental): Subjects in this arm will receive 6 monthly doses of 300 mg of lirentelimab (AK002) administered subcutaneously.
  Interventions: Drug: AK002
- SC 450 mg of lirentelimab (AK002) (Experimental): Subjects in this arm will receive 6 monthly doses of 450 mg of lirentelimab (AK002) administered subcutaneously.
  Interventions: Drug: AK002
- Placebo (Other): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AK002 — Lirentelimab (AK002) is a humanized non-fucosylated immunoglobulin G1(IgG1) monoclonal antibody directed against Siglec-8
  Other Names: Lirentelimab
  Arms: SC 150 mg of lirentelimab (AK002); SC 300 mg of lirentelimab (AK002); SC 450 mg of lirentelimab (AK002)
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy, safety, tolerability, and pharmacodynamic effect of subcutaneous lirentelimab (AK002), given monthly for 6 doses, in subjects with moderate to severe Eosinophilic Gastritis and/or Eosinophilic Duodenitis who have an inadequate response with, lost response to, or were intolerant to standard therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Male or female aged ≥18 and ≤80 years at the time of signing the informed consent for entry.
3. Baseline endoscopic biopsy with ≥30 eosinophils/hpf in at least 5 hpf in the stomach and/or ≥30 eosinophils/hpf in at least 3 hpf in the duodenum as determined by central histology assessment of biopsies collected during the screening EGD without any other significant cause for the eosinophilia.
4. Completion of at least 4 daily PRO questionnaires per week for a minimum of 3 weeks during screening.
5. A weekly average score of abdominal pain, nausea, or diarrhea ≥3 on the PRO questionnaire (score from 0-10) and a weekly average TSS of ≥10 for at least 2 weeks of screening.
6. Subjects with inadequate or loss of response to, or who were intolerant to standard therapies for EG and/or EoD, which could include PPI, antihistamines, systemic or topical corticosteroids, and/or diet, among others.
7. If subject is on preexisting dietary restrictions, willingness to maintain dietary restrictions throughout the study.
8. Willing and able to comply with all study procedures and visit schedule including follow-up visits.
9. Female subjects must be either post-menopausal for at least 1 year with FSH level >30 mIU/mL at screening or surgically sterile (tubal ligation, hysterectomy, or bilateral oophorectomy) for at least 3 months, or if of childbearing potential, have a negative pregnancy test and agree to use dual methods of contraception, or abstain from sexual activity from screening until the end of the study, or for 120 days following the last dose of study drug, whichever is longer. Male subjects with female partners of childbearing potential must agree to use a highly effective method of contraception from screening until the end of the study or for 120 days following the last dose of study drug, whichever is longer. All fertile men with female partners of childbearing potential should be instructed to contact the Investigator immediately if they suspect their partner might be pregnant (e.g., missed or late menstrual period) at any time during study participation.

Exclusion Criteria:

1. Use of systemic or topical corticosteroids exceeding the equivalent of 10 mg/day of prednisone within 4 weeks prior to the screening visit.
2. Change in the dose of corticosteroids (systemic or topical), PPI, leukotrienes, or diet therapy within 4 weeks prior to the screening visit.
3. Treatment with any immunosuppressive or immunomodulatory drugs that may interfere with the study within 12 weeks prior to the screening visit.
4. Prior exposure to AK002 or known hypersensitivity to any constituent of the study drug.
5. Active Heliobacter pylori (H. pylori) infection as confirmed by stool antigen test for H. pylori or identified in tissue biopsies obtained at screening EGD.
6. History of inflammatory bowel disease, celiac disease, achalasia, or esophageal surgery.
7. History of bleeding disorders and/or esophageal varices considered to be clinically significant by the Investigator.
8. Other significant gastric and/or duodenal eosinophilia or eosinophilic granulomatosis with polyangiitis (EGPA).
9. Confirmed diagnosis of hypereosinophilic syndrome (HES).
10. Women who are pregnant, breastfeeding, or planning to become pregnant while participating in the study.
11. Presence of an abnormal laboratory value considered to be clinically significant by the Investigator.
12. Any disease, condition (medical or surgical), or cardiac abnormality, which, in the opinion of the Investigator, would place the subject at increased risk.
13. History of malignancy, except carcinoma in situ, early-stage prostate cancer, or non-melanoma skin cancers. However, subjects with cancers that have been in remission for more than 5 years and are considered cured can be enrolled.
14. Treatment for a clinically significant helminthic parasitic infection within 6 months of screening.
15. Positive helminthic infection on Ova and Parasite (O&P) test.
16. Seropositive for Strongyloides stercoralis at screening.
17. Seropositive for HIV or hepatitis at screening except for vaccinated subjects or subjects with past but resolved hepatitis at screening.
18. Vaccination with live attenuated vaccines within 30 days prior to initiation of treatment in the study or expected during the treatment period. Vaccines authorized by FDA or other regulatory authority for the prevention of COVID-19 may be administered before, during, or after this protocol as per the label. The vaccine should not be administered within 7 days prior to and within 7 days after the administration of AK002 so that the side effects caused by either of the 2 medications can be more easily determined.
19. Participation in a concurrent interventional study with the last intervention occurring within 30 days prior to study drug administration (or 90 days or 5 half-lives, whichever is longer, for biologic products).
20. Known history of alcohol, drug, or other substance abuse or dependence that is considered by the Investigator to be ongoing and clinically significant.
21. Any other reason that in the opinion of the Investigator or the Medical Monitor makes the subject unsuitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Proportion of Responders as determined by gastric or duodenal tissue eosinophil counts. | At Week 24
  A responder is a subject achieving the following peak eosinophil counts: eosinophil count ≤4 cells per hpf in 5 gastric hpf and/or eosinophil count ≤15 cells per hpf in 3 duodenal hpf
Mean absolute change in 6 symptom total symptom score (TSS: abdominal pain, nausea, abdominal cramping, loss of appetite, fullness before finishing a meal, and bloating ) as measured by the PRO questionnaire (score from 0 none - 10 worst) | Baseline to Weeks 23 - 24

SECONDARY OUTCOMES:
Percent change in tissue eosinophils | Baseline to Week 24
Number of treatment responders as defined by >30% improvement in symptoms and mean eosinophil count ≤4 cells/hpf in 5 gastric hpf and/or mean eosinophil count ≤15 cells/hpf in 3 duodenal hpf. | Baseline to Weeks 23-24 and at Week 24, respectively.
Proportion of subjects achieving mean eosinophil count ≤1 cell/hpf in 5 highest gastric hpf and mean eosinophil count ≤1 cell/hpf in 3 highest duodenal hpf | At Week 24
Proportion of subjects who show ≥50% reduction in TSS | Baseline to Weeks 23-24
Proportion of subjects who show ≥70% reduction in TSS | Baseline to Weeks 23-24
Change in weekly TSS over time | Baseline to Weeks 23-24

CONTACTS AND LOCATIONS:
Overall Officials: Craig Paterson, MD, Study Director — Allakos Inc.
Locations (73):
- United States (73):
  - Allakos Investigational Site, Birmingham, Alabama
  - Allakos Investigational Site, Gilbert, Arizona
  - Allakos Investigational Site, Phoenix, Arizona
  - Allakos Investigational Site, Scottsdale, Arizona
  - Allakos Investigational Site, Chula Vista, California
  - Allakos Investigational Site, Long Beach, California
  - Allakos Investigational Site, Ventura, California
  - Allakos Investigational Site, Walnut Creek, California
  - Allakos Investigational Site, Bristol, Connecticut
  - Allakos Investigational Site, Brandon, Florida
  - Allakos Investigational Site, Edgewater, Florida
  - Allakos Investigational Site, Jacksonville, Florida
  - Allakos Investigational Site, Kissimmee, Florida
  - Allakos Investigational Site, Miami, Florida
  - Allakos Investigational Site, New Port Richey, Florida
  - Allakos Investigational Site, Ponte Vedra, Florida
  - Allakos Investigational Site, Sunrise, Florida
  - Allakos Investigational Site, Tampa, Florida
  - Allakos Investigational Site, Atlanta, Georgia
  - Allakos Investigational Site, Sandy Springs, Georgia
  - Allakos Investigational Site, Chicago, Illinois
  - Allakos Investigational Site, Iowa City, Iowa
  - Allakos Investigational Site, Kansas City, Kansas
  - Allakos Investigational Site, Crowley, Louisiana
  - Allakos Investigational Site, Shreveport, Louisiana
  - Allakos Investigational Site, Glen Burnie, Maryland
  - Allakos Investigational Site, Boston, Massachusetts
  - Allakos Investigational Site, Ann Arbor, Michigan
  - Allakos Investigational Site, Wyoming, Michigan
  - Allakos Investigational Site, Rochester, Minnesota
  - Allakos Investigational Site, Bay Saint Louis, Mississippi
  - Allakos Investigational Site, Flowood, Mississippi
  - Allakos Investigational Site, Kansas City, Missouri
  - Allakos Investigational Site, Kalispell, Montana
  - Allakos Investigational Site, Reno, Nevada
  - Allakos Investigational Site, Lebanon, New Hampshire
  - Allakos Investigational Site, Florham Park, New Jersey
  - Allakos Investigational Site, Freehold, New Jersey
  - Allakos Investigational Site, Great Neck, New York
  - Allakos Investigational Site, New York, New York
  - Allakos Investigational Site, Chapel Hill, North Carolina
  - Allakos Investigational Site, Charlotte, North Carolina
  - Allakos Investigational Site, Concord, North Carolina
  - Allakos Investigational Site, Durham, North Carolina
  - Allakos Investigational Site, Raleigh, North Carolina
  - Allakos Investigational Site, Winston-Salem, North Carolina
  - Allakos Investigational Site, Cincinnati, Ohio
  - Allakos Investigational Site, Columbus, Ohio
  - Allakos Investigational Site, Dayton, Ohio
  - Allakos Investigational Site, Mentor, Ohio
  - Allakos Investigational Site, Springboro, Ohio
  - Allakos Investigational Site, Westlake, Ohio
  - Allakos Investigational Site, Oklahoma City, Oklahoma
  - Allakos Investigational Site, Philadelphia, Pennsylvania
  - Allakos Investigational Site, Greenwood, South Carolina
  - Allakos Investigational Site, Chattanooga, Tennessee
  - Allakos Investigational Site, Germantown, Tennessee
  - Allakos Investigational Site, Hixson, Tennessee
  - Allakos Investigational Site, Nashville, Tennessee
  - Allakos Investigational Site, Austin, Texas
  - Allakos Investigational Site, El Paso, Texas
  - Allakos Investigational Site, Fort Worth, Texas
  - Allakos Investigational Site, Lubbock, Texas
  - Allakos Investigational Site, San Antonio, Texas
  - Allakos Investigational Site, Southlake, Texas
  - Allakos Investigational Site, Webster, Texas
  - Allakos Investigational Site, Wichita Falls, Texas
  - Allakos Investigational Site, Ogden, Utah
  - Allakos Investigational Site, Riverton, Utah
  - Allakos Investigational Site, Salt Lake City, Utah
  - Allakos Investigational Site, Sandy City, Utah
  - Allakos Investigational Site, Fairfax, Virginia
  - Allakos Investigational Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No